CLINICAL TRIAL: NCT02989350
Title: Efficacy of Lactobacillus Reuteri DSM 17938 for the Treatment of Acute Gastroenteritis in Children: Randomised Controlled Trial
Brief Title: Efficacy of Lactobacillus Reuteri DSM 17938 for the Treatment of Acute Gastroenteritis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szpital im. Św. Jadwigi Śląskiej (Other)
Responsible Party: Principal Investigator, Henryk Szymański, MD PhD, Szpital im. Św. Jadwigi Śląskiej
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1/2016
Record Dates: First submitted 2016-12-01; First posted 2016-12-12 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Acute Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus reuteri DSM 17938 (Active Comparator): 2 x 10(8) CFU. Both L reuteri DSM 17938 and placebo will be taken orally, twice daily 5 drops, for consecutive 5 days.
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938
- Placebo (Placebo Comparator): Placebo consists of an identical formulation, except active substance.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17938 — Lactobacillus reuteri DSM 17938 vs Placebo
  Arms: Lactobacillus reuteri DSM 17938
Dietary Supplement: Placebo — Lactobacillus reuteri DSM 17938 vs Placebo
  Arms: Placebo

SUMMARY:
Acute gastroenteritis (AGE) is one of the most common diseases among children. Oral rehydration therapy is the key treatment. According to the 2014 guidelines developed by the ESPGHAN probiotics may be considered in the management of children with AGE in addition to rehydration therapy. Considering that evidence on L reuteri remains limited, the investigators aim to assess the efficacy of L reuteri DSM 17938 for the treatment of AGE in children. Children vaccinated and not vaccinated against rotavirus will be evaluated separately.

Two independent reports (rotavirus-vaccinated and non-vaccinated children) are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Acute gastroenteritis (AGE) defined as a change in stool consistency to loose or liquid form (according to the Bristol Stool Form (BSF) scale or in the case of infants, the Amsterdam Stool Form (ASF) scale) and/or an increase in the frequency of evacuations (typically ≥3 in 24 h), lasting for no longer than 5 days.
2. Age: older than 1 month and younger than 60 months.
3. A caregiver must provide written informed consent.

Exclusion Criteria:

1. Use of antibiotics within two weeks prior to enrolment.
2. Use of gelatine tannate, diosmectite, probiotics, racecadotril, or zinc (including zinc containing ORS) within a week prior to enrolment (a single dose is allowed).
3. Breast feeding (>50%)
4. Chronic diarrhoeal gastrointestinal disease (e.g., inflammatory bowel disease, cystic fibrosis, coeliac disease, food allergy)
5. Immunodeficiency
6. Malnutrition (weight/height/length under 3rd percentile) (WHO Child Growth Standards will be used)

Ages: 2 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | 8 days
  (measured in hours) - time until the normalisation of stool consistency according to the Bristol Stool Form Scale(BSF) or Amsterdam Infant Stool Scale (ASF) - (in BSF scale, numbers 1, 2, 3, 4 and 5; in ASF scale, letters B or C), or the time until the normalisation of the number of stools (compared with the period before the onset of diarrhoea).and the presence of normal stools for 48 h.

SECONDARY OUTCOMES:
Need for intravenous rehydration | 8 days
  Number of patients in each group requiring intravenous rehydration
Duration of intravenous rehydration | 8 days
Need for hospitalisation of outpatients | 8 days
  Number of patients enrolled as outpatient requiring hospitalisation - based on medical assesment
Number of watery stools per day | 8 days
Vomiting | 8 days
  Number of participants with vomits and number of vomits per day
Recurrence of diarrhoea (in 48 hours after intervention) | 48 hours
  Number of patients in which diarrhoea recur after initial recovery in 48 hours
Severity of diarrhoea according to Vesikari scale | 8 days
Use of concomitant medications | 8 days
Adverse events | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Henryk Szymański, MD PhD, Principal Investigator — Szpital im.Świętej Jadwigi Śląskiej, Trzebnica, Poland
Locations (1):
- Szpiatal im.Świętej Jadwigi Śląskiej, Trzebnica, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Szymanski H, Szajewska H. Efficacy of Lactobacillus Reuteri DSM 17938 for the Treatment of Acute Gastroenteritis in Children: Protocol of a Randomized Controlled Trial. JMIR Res Protoc. 2017 Aug 23;6(8):e164. doi: 10.2196/resprot.7924. PMID 28835355
- See also: published protocol — http://www.researchprotocols.org/2017/8/e164/